CLINICAL TRIAL: NCT06911151
Title: Innovative Footwear for People Experiencing Foot Drop; a Feasibility Study
Brief Title: Innovative Shoe for People With Foot Drop
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Margaret University (Other)
Responsible Party: Principal Investigator, Marietta van der Linden, Professor, Queen Margaret University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIHR207749; NIHR207749 (Other Grant/Funding Number: NIHR)
Record Dates: First submitted 2025-03-21; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Foot Drop
Keywords: foot drop; gait; trips and falls; footwear; walking disability
MeSH Terms: conditions — Peroneal Neuropathies; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: pre- post single group design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- innovative footwear (Experimental): The Edinburgh-based Health Design Collective (HDC), led by three physiotherapists and one podiatrist and supported by people with lived experience, have designed footwear that incorporates the support needed to reduce foot drop. This footwear includes 'Smartstrap Technology' - integrated elastic straps that help to hold the foot in a good position when walking. The footwear does not require any additional devices and people who have tested it find that the footwear makes their walking easier, while also being usable, comfortable, and unobtrusive.
  Interventions: Device: innovative footwear

INTERVENTIONS:
Device: innovative footwear — HDC shoe

SUMMARY:
People with foot drop have an increased risk of tripping and falling, and this makes walking more difficult. Our colleagues at the Health Design Collective (HDC) have developed a shoe that aims to make it easier for people with foot drop to walk. People who have tested a prototype of the shoe, have told us that it makes their walking easier, but is also comfortable and unobtrusive. However, the investigators need more scientific evidence that this shoe helps reduce foot drop and improves walking in people with foot drop. The purpose of this small study, with only 15 participants, is to lay the foundations to design and carry out a bigger study. participants have been asked to take part if they are aged 18+ years and have experienced foot drop in the past 6 months or more. To be able to take part in this study participants need to be able to walk for 2 minutes without stopping (with or without their normal walking aid) and have sufficient movement in their ankle to use the shoe. Unfortunately, if the participant has severe swelling of their legs, deep vein thrombosis, or severe problems with the skin on their feet, they will not be able to take part in this study. If the participant agrees to take part, they will be fitted with a pair of the new shoes and asked to try them out for a period of 6 weeks. They will continue to wear any orthotics/ankle foot orthotics or other aids that they are currently using. Before and during these six weeks the investigators will ask the participant to wear a small device that measures their physical activity. Just before and after these 6 weeks the investigators will invite the participant to Queen Margaret University for some walking tests with the new shoes. The investigators will also ask the participant to complete several questionnaires which they can do at home. After the 6-week shoe testing period the investigators will invite the participant for an interview, either in person or remotely, during which they can tell the researchers their thoughts about the new shoe. Participants will be asked to travel to Queen Margaret University, Musselburgh and all of their travel expenses to and from the university will be reimbursed. The study involves testing a new shoe which participants might find uncomfortable and take some time to get used to. The investigators will support participants throughout 6 weeks testing period to make sure that they are safe and free of pain when using the shoes. If participants experience any issues related to the shoes, they should stop wearing them and contact the investigators. The two study assessments will involve several walking tests that participants may find tiring. People who have tested an early prototype of the shoe, have told the research team that it makes their walking easier, but is also comfortable and unobtrusive. However, it is possible participants will not experience these benefits. The investigators hope this study also helps people in the future to find out more about how this research can develop the shoes and how it impacts people affected by foot drop. If participants find them useful, they can keep the shoes after taking part in the study. If they are interested in taking part in this study after reading this information sheet, please contact the researcher to discuss the study and ask any questions. If participants decide to take part, they will be asked to complete a paper or electronic consent form. If they are happy to sign the consent form, the research team will send them a short survey with a couple of questions such as their age, shoe size, health condition, and how long they have experienced foot drop. This will allow the research team to order shoes in the correct size for the participant. Once the study period starts, the participant will record any falls they have had over a period of 6 weeks in either a paper or electronic diary, whichever they prefer. It is valuable for the General Practitioner (GP), orthotist and podiatrist, to know who is taking part in research. If the participant has given the investigators consent to do so, the research team will inform the participants GP, orthotist and podiatrist that the participant is taking part in the study.

In addition, the participant will be sent a small, lightweight activity monitor (picture below) and asked to wear it by attaching it to their leg for a period of 7 days. This monitor records how many steps that are taken each day and how fast the person is walking. The participant will be asked to wear the monitor whilst sleeping, if possible, but they will need to remove it for bathing and swimming. After a period of about 6 weeks, the investigators will invite the participant to Queen Margaret University, Musselburgh to fit them with a pair of HDC shoes. If English is the 2nd language, the person may bring a translator if they wish. Any travel expenses to and from the University will be reimbursed.

DETAILED DESCRIPTION:
The investigators will ask the participant to carry out two different types of walking tests. Both tests will be repeated twice: 1) with new shoes but with no tension (standard shoes) 2) with the new shoes applying tension using a special strap which is designed to reduce foot drop. participants are allowed to rest between each test for as long as they need and may use their usual walking aids. The first test involves walking around two cones about 10 meters apart for a maximum of 2 minutes without stopping.

For the second type of walking test, the investigators will need to attach small reflective balls (markers) to their legs and pelvis using skin-friendly sticky tape (see picture below). Using special cameras that only see the reflective markers, the researchers can create a very detailed and accurate measurement of how their legs move when they walk. For this walking test, researchers will ask participants to walk about 6 meters, six times: three times using the shoes with no tension, and three times in the shoes with the tension applied to the affected foot. Participants can walk at a speed that is comfortable to them and can stop and rest whenever they wish. Investigators will ask participants to complete two questionnaires, one about how their health condition affects their quality of life, and the other one about which clinical services (e.g. GP, physiotherapy) they have used in the past 6 weeks. participants can complete these at home before their visit or after the walking tests, either in paper or electronic format, whichever they prefer. It should take no more than half an hour to complete these questionnaires.

Investigators will also ask participants to rate their our ability to carry out up to five daily activities that are important to them (e.g., walking upstairs, shopping, doing housework), on a scale of 1 (can't do it activity) to 10 (I have no problem at all doing this activity).

After the first visit

Researchers will ask participants to use the new shoe with the special strap at home for a duration of 6 weeks. During the first week, they will be asked to follow a safety and footwear adaptation protocol which will help them get used to the shoes. For the following five weeks, they are free to use the shoes whenever they wish. During the 6 weeks between visits, investigators will ask participants to complete an electronic or paper diary recording their use of the shoes and any specific challenges/feedback and whether they had a fall. If participants have any questions or need any help to complete the diary or with wearing the shoes, they can contact the researcher at any point.

A week before the second scheduled visit, researchers will ask participants to wear the activity monitor on their leg again for a period of 7 days. The process for the second visit will be the same as the first visit, except for a short additional footwear survey to find out the opinions about the shoes. Interviews will be conducted in person or remotely, depending on the preference. The remote interviews will be carried out online or by telephone. All interviews will be recorded using a digitally encrypted audio recorder. Interviews will be carried out to find out the views and perspectives relating to the use of the new shoes. participants will be asked about their positive and negative experiences or impacts and thoughts on the ongoing use of new shoes. It is not thought that there are any disadvantages; however, it is important that participants are careful when they start to use the new shoes. They will need to become accustomed to the shoe, which may take up to 1 week. Investigators will support participants and help by giving a safety protocol to follow. If there are any concerns at any time, people are advised to immediately stop wearing the shoes and contact the researcher to discuss. The researcher's contact details are provided in the diary, please also record all safety concerns in the diary. Key areas of safety concerns are as follows:

When wearing the shoe, has the participant had any falls or near falls?

When the participant wears the shoe, do they experience any pain?

After wearing the shoe, do they notice any areas of skin redness or skin breakdown?

As previously explained, people can withdraw from the study at any point, without having to give a reason.

At the end of the study, people can keep the pair of new shoes at no cost if they have found them useful. If participants would like to receive a lay summary of the study findings, researchers can send this once they have finished analysing the data.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18+ years
* Individuals experiencing foot drop as diagnosed by a health professional due to any health condition for 6 months or more
* the ability to walk at least 6 metres (with or without walking aid) at their own pace
* with capacity to consent
* Those with English as a 2nd language may bring a translator.

Exclusion Criteria:

* impaired cognitive function (as assessed in the initial phone call using elements of the Abbreviated Mental Test Score27) and questions that will assess the potential participant's understanding of the research protocol);
* inability to achieve minimum 10 degrees ankle flexion;
* lymphoedema of lower limbs/ deep vein thrombosis in the last 6 months;
* any change in medication/treatment in the last 3 months that may cause a change in walking experience;
* existing pressure areas at risk of, or active skin breakdown in areas that will make contact with the inner of the shoe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
daily use of HDC footwear | from baseline (t0) , every day to the end of the intervention period at 6 weeks
  Baseline (t0): Participants are given a paper or electronic diary at baseline, in which they record for each day during the 6 week intervention period how often and how long they used the new footwear (HDC shoe). They will also record any adverse events related to wearing the HDC shoe

SECONDARY OUTCOMES:
Timed 2 minute walk test | at baseline (t0)
  At baseline (t0): walking will be assessed through the 2 minute walking test at baseline (t0) . Participants will be asked to walk up and down the motion analysis laboratory around 2 cones, placed 10 metres apart, for a duration of 2 minutes. They will be instructed to cover as much distance as possible in a safe manner within a two minute duration without stopping to rest. Participants will be allowed to use their normal walking aids.
Timed 2 minute walk test | after 6 weeks with the intervention (t1)
  After 6 weeks with the intervention (t1) walking will be assessed through the 2 minute walking test. Participants will be asked to walk up and down the motion analysis laboratory around 2 cones, placed 10 metres apart, for a duration of 2 minutes. They will be instructed to cover as much distance as possible in a safe manner within a two minute duration without stopping to rest. Participants will be allowed to use their normal walking aids.
Canadian Occupational Performance Measure | at baseline (t0)
  At baseline (t0) participants will complete the COPM wh9ch is a semi-structured interview, ratings from 1 to 10, higher scores indicate higher perceived improvement in function
Canadian Occupational Performance Measure | at the end of the intervention period at 6 weeks (t1)
  At the end of the intervention period at 6 weeks (t1) participants will complete the COPM which is a semi-structured interview, ratings from 1 to 10, higher scores indicate higher perceived improvement in function
Weekly step count | seven days before baseline (t0)
  Participants will wear the activity monitor for the seven days before baseline, measured using an ActivPal activity monitor
Weekly step count | at week 5, which is one week before the end of the 6 week intervention period (t1)
  Participants will wear the activity monitor for seven days measured using an ActivPal activity monitor
Gait analysis | baseline (t0)
  At baseline (t0) Gait analysis with the vicon motion analysis. Computerised three domensional gait analysis will be used to measure lower limb kinematics, and specifically joint angles between the foot and the lower limb segment to measure dorsiflexion movement in the sagittal plane.
Gait analysis | after the 6 week intervention period, at 6 weeks (t1)
  After the 6 week intervention period at 6 weeks (t1), Gait analysis with the vicon motion analysis. Computerised three domensional gait analysis will be used to measure lower limb kinematics, and specifically joint angles between the foot and the lower limb segment to measure dorsiflexion movement in the sagittal plane.
Falls | starting at day 1, for 6 weeks prior to baseline (t0)
  For 6 weeks prior to baseline (t0), The participants will be asked to record any trips and / or falls that they have in a falls diary.
Falls | from baseline (t0) until the end of the intervention period at 6 weeks (t1)
  During the 6 week intervention period, from baseline (t0) until the end of the 6 week intervention period at 6 weeks (t1),The participants will be asked to record any trips and / or falls that they have in a falls diary.
Euro-Qol EQ-5D | baseline (t0)
  At baseline (t0), Quality of life survey
Euro-Qol EQ-5D | After the 6 week intervention period at 6 weeks (t1)
  After the 6 week intervention period at 6 weeks (t1), Quality of life survey
Footwear Survey | After the 6 week intervention period at 6 weeks (t1)
  After the 6 week intervention period at 6 weeks (t1), A survey to determine the participants thoughts and opinions on the footwear
Health evaluation survey | baseline (t0)
  At baseline (t0), Health evaluation survey to determine the financial implications of the burden of foot drop
Health evaluation survey | at the end of the 6 week intervention period at 6 weeks (t1)
  At the end of the 6 week intervention period at 6 weeks (t1), Health evaluation survey to determine the financial implications of the burden of foot drop

OTHER OUTCOMES:
Qualitative Interviews | At three weeks after the intervention period (t1), at 9 weeks
  at three weeks after the end of the intervention period, Interviews will be conducted from a constructivist phenomenological perspective, aiming to explore the views and perspectives of the participants relating to the use of the new footwear.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Margaret University, Edinburgh, Lothian, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
anonymous data may be shared on request from other researchers

REFERENCES:
- [Background] Kadaba MP, Ramakrishnan HK, Wootten ME. Measurement of lower extremity kinematics during level walking. J Orthop Res. 1990 May;8(3):383-92. doi: 10.1002/jor.1100080310. PMID 2324857
- [Background] Bulley C, Shiels J, Wilkie K, Salisbury L. User experiences, preferences and choices relating to functional electrical stimulation and ankle foot orthoses for foot-drop after stroke. Physiotherapy. 2011 Sep;97(3):226-33. doi: 10.1016/j.physio.2010.11.001. Epub 2011 Feb 2. PMID 21820541